CLINICAL TRIAL: NCT04038437
Title: A Phase 1b Trial of CPX-351 Lower Intensity Therapy (LIT) Plus Venetoclax as First Line Treatment for Subjects With AML Who Are Unfit for Intensive Chemotherapy
Brief Title: A Trial of CPX-351 Lower Intensity Therapy (LIT) Plus Venetoclax as First Line Treatment for Subjects With AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX351-103
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: CPX-351; Vyxeos; Venetoclax; Unfit
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPX-351 and Venetoclax (Experimental): CPX-351 and Venetoclax will be administered over 28 day cycles
  Interventions: Drug: CPX-351; Drug: Venetoclax

INTERVENTIONS:
Drug: CPX-351 — CPX-351 will be administered on Days 1 and 3 of each cycle
  Other Names: Vyxeos
Drug: Venetoclax — Venetoclax will be adminstered on Days 2 to 21 of each cycle
  Other Names: Venclexta

SUMMARY:
Study CPX351-103 is an open-label, multicenter, phase 1b, safety and PK study to determine the MTD of the combination of CPX 351 and venetoclax when administered to subjects with newly diagnosed AML who are unfit for intensive chemotherapy (ICT) and to determine the recommended phase 2 dose (RP2D) for the Expansion Phase. This study will comprise 2 phases: a Dose Exploration Phase (Part 1) and an Expansion Phase (Part 2), in which all subjects will receive a combination of CPX-351 and venetoclax.

ELIGIBILITY:
Inclusion Criteria:

• Subject must have newly diagnosed AML with histological confirmation by World Health Organization (WHO) criteria.

Definition of subjects who are unfit for ICT:

• Each subject must meet the following criteria characterizing him / her as unfit to receive ICT prior to the first day of therapy to be enrolled in the study:

* ≥ 75 years of age OR
* ≥ 18 to 74 years of age and fulfilling at least 1 criteria associated with lack of fitness for ICT as follows:

  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 to 3;
  * Cardiac history of Congestive Heart Failure (CHF) requiring treatment or left ventricular ejection fraction (LVEF) ≤ 50%.
  * Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) ≤ 65% or Forced Expiratory Volume in 1 second (FEV1) ≤ 65%;
  * Creatinine clearance (CrCl) ≥ 30 mL/min to < 45 mL/min calculated by the Cockcroft-Gault formula;
  * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × Upper Limit of Normal (ULN);
  * Other comorbidity that the physician judges to be incompatible with conventional intensive chemotherapy which must be reviewed and approved by the study medical monitor before study enrollment.

In addition, all subjects must meet the following criteria:

* If the subject is ≥ 75 years of age, then ECOG Performance Status must be 0-2.
* Subject must have adequate renal function as demonstrated by a CrCl ≥ 30 mL/min (calculated by the Cockcroft Gault formula or measured by 24-hour urine collection).
* Subject must have adequate liver function as demonstrated by:

  * Aspartate aminotransferase (AST) ≤ 3.0 × ULN*
  * Alanine aminotransferase (ALT) ≤ 3.0 × ULN*
  * Bilirubin ≤ 1.5 × ULN (subjects who are < 75 years of age may have bilirubin of ≤ 3.0 × ULN)* *Unless considered to be due to leukemic organ involvement.
* Female subjects must be either postmenopausal defined as:

  * Age > 55 years with no menses for ≥ 2 years without an alternative medical cause.
  * OR
  * Age ≤ 55 years with no menses for ≥ 12 months without an alternative medical cause AND a follicle-stimulating hormone level > 40 IU/L;
  * OR
  * Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy); OR
* A woman of childbearing potential practicing at least 1 protocol specified method of birth control starting at Study Day 1 through at least 6 months after the last dose of study treatment.
* A woman of childbearing potential must have negative results for pregnancy test performed:

  * At Pretreatment with a serum sample obtained within 28 days prior to the first study treatment administration, and
  * Prior to dosing with urine sample obtained on Cycle 1 Day 1, if it has been > 7 days since obtaining the serum pregnancy test results.
  * Subjects with borderline pregnancy tests at Pretreatment must have a serum pregnancy test ≥ 3 days later to document continued lack of a positive result.
* Male subjects who are sexually active, must agree, from Study Day 1 through at least 6 months after the last dose of study treatment, to practice protocol specified methods of contraception. Male subjects must agree to refrain from sperm donation from initial study treatment administration through at least 6 months after the last dose of study treatment.
* Subject must have a white blood cell count ≤ 25 × 10^9/L. (Note: subjects who have undergone hydroxyurea administration or leukapheresis for therapeutic cytoreduction will be considered eligible).

Exclusion Criteria:

* Subject has ECOG Performance Status > 3, regardless of age.
* Subject has known Human Immunodeficiency Virus (HIV) infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax). HIV testing will be performed at Pretreatment, if required per local guidelines or institutional standards.
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as determined by the specified dose exploration | Up to 36 months
  The Recommended Phase 2 Dose (RP2D) as determined by an assessment of all safety data from the Dose Exploration Phase.
Incidence of Adverse Events (AE) and Dose Limiting Toxicities (DLT) | Up to 36 months
  The safety and tolerability of CPX-351 and venetoclax when given in combination based on the incidence of AEs and DLTs

SECONDARY OUTCOMES:
Proportion of subjects who have achieved CR, CRi, PR, and CRc (CR + CRi) | Up to 36 months
  Proportion of subjects who have achieved CR, CRi, PR, and CRc (CR + CRi) at any time while receiving study treatment.
Proportion of subjects who have achieved ORR | Up to 36 months
  Proportion of subjects who have achieved ORR, defined as best response (CR + CRi + PR) at any time while receiving study treatment.
Proportion of subjects who have achieved CR / CRi with MRD status | Up to 36 months
  Proportion of subjects who have achieved CR / CRi with MRD status (negative / positive) at any time while receiving study treatment.
AUCtau | Exploration: Cycle 1, Days 1 and 3: predose, 45 and 90 minutes (min), 4, 6, and 8 hours(hr); Days 2 and 4: 24 hr; Day 5: 48 hr; Cycle 2 Day 3: predose, 45 and 90 min, 4, 5, 6, and 8 hr; Day 4: 24 hr; Day 5: 48 hr (each cycle is 28-49 days)
  Area under the plasma concentration time curve from time 0 to the time of the next dosing during a 48 hour interval at the steady-state of CPX-351 PK
Maximum Plasma Concentration (Cmax) | Exploration:Cycle 1,Days 1 and 3:predose,45 and 90 minutes(min),4,6, and 8 hours (hr); Days 2 and 4:24 hr; Day 5:48 hr; Day 7:96 hr, Day 9:144 hr; Cycle 2 Day 3:predose,45 and 90 min,4,5,6, and 8 hr; Day 4:24 hr; Day 5:48 hr (each cycle is 28-49 days)
Time to Cmax (Tmax) | Exploration:Cycle 1,Days 1 and 3:predose,45 and 90 minutes(min),4,6, and 8 hours (hr); Days 2 and 4:24 hr; Day 5:48 hr; Day 7:96 hr, Day 9:144 hr; Cycle 2 Day 3:predose,45 and 90 min,4,5,6, and 8 hr; Day 4:24 hr; Day 5:48 hr (each cycle is 28-49 days)
Apparent Terminal Elimination Half-Life (t½) | Exploration:Cycle 1,Days 1 and 3:predose,45 and 90 minutes(min),4,6, and 8 hours (hr); Days 2 and 4:24 hr; Day 5:48 hr; Day 7:96 hr, Day 9:144 hr; Cycle 2 Day 3:predose,45 and 90 min,4,5,6, and 8 hr; Day 4:24 hr; Day 5:48 hr (each cycle is 28-49 days)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Blood & Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana Farber/ Brigham & Women's Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Uy GL, Pullarkat V, Baratam P, Stuart RK, Walter RB, Winer ES, Wang Q, Faderl S, Chakravarthy D, Menno D, Cheung RS, Lin TL. Lower-intensity CPX-351 plus venetoclax induction for adults with newly diagnosed AML unfit for intensive chemotherapy. Blood Adv. 2024 Dec 24;8(24):6248-6256. doi: 10.1182/bloodadvances.2024013687. PMID 39418644